CLINICAL TRIAL: NCT02142621
Title: Pilot N-of-1 Multiple Crossover Randomized Trial of Gastric and Transpyloric Feeds in Infants With Severe Bronchopulmonary Dysplasia
Brief Title: Transpyloric Feeding in Severe Bronchopulmonary Dysplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14-010924
Record Dates: First submitted 2014-05-15; First posted 2014-05-20 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- transpyloric tube feeds (Active Comparator): Continuous transpyloric tube feeds administered through an oral/nasal feeding tube.
  Interventions: Other: transpyloric feeding
- gastric tube feeds (Active Comparator): Continuous gastric tube feeds administered through an oral/nasal feeding tube.
  Interventions: Other: gastric feeding

INTERVENTIONS:
Other: transpyloric feeding
  Arms: transpyloric tube feeds
Other: gastric feeding
  Arms: gastric tube feeds

SUMMARY:
Bronchopulmonary dysplasia (BPD) is the most common complication of extreme preterm birth. It impacts 10,000-15,000 infants in the US annually, including approximately 50% of infants with birth weight < 1000g. BPD is associated with multiple long-term adverse outcomes including chronic cardiopulmonary and neurodevelopmental impairments. Infants with severe BPD, defined as a need for ≥ 30% inspired oxygen and/or mechanical respiratory support at 36 weeks postmenstrual age (PMA), suffer the greatest burden of these chronic sequelae. Recurrent episodes of hypoxemia and prolonged exposure to supplemental oxygen are linked to the development of these impairments. Gastroesophageal reflux (GER) contributes to these mechanisms by exacerbating pulmonary inflammation and inducing bronchospasm. Unfortunately, clinically available methods to diagnose GER in infants are unreliable. Moreover, acid suppressive agents are both ineffective and carry high risk of serious life-threatening morbidity. Simple transpyloric feeding has promise, but has not been evaluated in BPD.

This study will pilot N-of-1 trials to assess whether transpyloric feeds reduce airway complications of GER and and whether this methodology can aid in identifying individual infants with severe BPD who are likely to benefit from prolonged use of transpyloric feeds.

Aim 1. To determine for each enrolled infant with severe BPD whether transpyloric compared to gastric feeds reduce the number of daily intermittent hypoxemic events (primary outcome) and improve a validated BPD severity score (secondary outcome).

The investigators hypothesize that 80% percent of enrolled infants will have significantly fewer daily intermittent hypoxemic events with transpyloric compared to gastric feeds and will have this feeding method formally recommended.

Aim 2. To pool results from multiple N-of-1 trials to determine whether transpyloric compared to gastric feeds reduce airway complications of GER in infants with severe BPD.

The investigators hypothesize that transpyloric compared to gastric feeds will be associated overall with a 15% reduction in number of daily intermittent hypoxemic events.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≤ 32 weeks
* Severe BPD (FiO2 ≥ 30% and/or mechanical ventilation or non-invasive positive pressure respiratory support at the time of enrollment)
* Post menstrual age of 36-45 6/7 weeks at enrollment
* Parent and/or guardian permission (informed consent)

Exclusion Criteria:

* Prior intolerance to transpyloric feeds
* History of surgical anti-reflux procedure
* Congenital heart disease (not including patent ductus arterioles and hemodynamically insignificant ventricular septal defect or atrial septal defect)
* Structural abnormalities of the upper airway, lungs, or chest wall
* Other congenital malformations or syndromes that adversely affect life expectancy or cardio-pulmonary development
* Parent, guardian, or subject who, in the opinion of the investigators, are unlikely to participate for the duration of the study

Ages: 4 Weeks to 24 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
Change in transient intermittent hypoxemic events every 4 days | 4 days
  transient hypoxemic events is defined for the purposes of this study as an oxygen saturation < 80% for ≥ 10 seconds and < 3 minutes recorded by continuous pulse oximetry.

CONTACTS AND LOCATIONS:
Overall Officials: Haresh Kirpalani, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Jensen EA, Zhang H, Feng R, Dysart K, Nilan K, Munson DA, Kirpalani H. Individualising care in severe bronchopulmonary dysplasia: a series of N-of-1 trials comparing transpyloric and gastric feeding. Arch Dis Child Fetal Neonatal Ed. 2020 Jul;105(4):399-404. doi: 10.1136/archdischild-2019-317148. Epub 2019 Nov 4. PMID 31685527